CLINICAL TRIAL: NCT03293225
Title: A Randomized Open Labeled Trial to Compare the Efficacy of Antihistamine Dosing-up and add-on Treatment With H2-receptor Antagonist in Patients With Chronic Urticaria
Brief Title: Efficacy of Antihistamine Dosing-up and add-on Treatment With H2-receptor Antagonist
Acronym: OPEhRA
Status: Completed | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ye Youngmin, professor, Department alleric internal medicine, Ajou University School of Medicine
Other Study IDs: AJIRB-MED-OBS-17-173
Record Dates: First submitted 2017-09-11; First posted 2017-09-26 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Chronic Urticaria
Keywords: cu
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- add H2RA: Add antihistamines to standard drug therapy
- change ns-H1RA: Change to ns-H1RA in standard medication
- ns-H1RA(3-4 tabs): Standard treatment with ns-H1RA 4X dose
- ns-H1RA(3-4kinds): Use of NS 4 kinds for standard treatment

SUMMARY:
A randomized open labeled trial to compare the efficacy of antihistamine dosing-up and add-on treatment with H2-receptor antagonist in patients with chronic urticaria

DETAILED DESCRIPTION:
* For four weeks
* After the researcher confirms the selection / exclusion criteria on the baseline, the UAS, K-UCT, and CU-QoL are created and randomized from the subject.
* Receive UAS, K-UCT, and CU-QoL from the subject during the last visit to assess safety

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and adults over 12 years
* Clinical diagnosis of chronic urticaria due to wheal reaction, itching, angioedema over 6 weeks
* Antihistamine 2 or 2 kinds of treatment for more than 2 weeks even if the symptoms are not controlled
* Those who do not have other chronic skin diseases

Exclusion Criteria:

* None

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic urticaria in Ajou University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Number of evaluation after 4 weeks treatment by a investigator | 4 weeks
  0-no effective, 1-ineffective, 2-effective, 3-no symptoms

SECONDARY OUTCOMES:
Peripheral blood eosinophil count | 4 weeks
  in percentage
Number of evaluation as assessed by questionnaire | 4 weeks
  Sleepiness, dryness, dysuria
Number of urticaria control by K-UCT | 4 weeks
  Before and after treatment
Number of urticaria symptom by UAS | 4 weeks
  Urticaria activity score
Quality of life of chronic urticaria by CU-QoL | 4 weeks
  Quality of life questionnaire for patients with chronic urticaria
Number of Patient-controlled urticaria by VAS | 4 weeks
  evaluation of Patient-controlled urticaria
Number of patients using emergency medication | 4 weeks
  Emergency drug frequency in patients with chronic urticaria
Comparison of Serum total IgE | 4 weeks
  Comparison each group in treatment activity
Number of physiological parameter | 4 weeks
  weight gain in kilograms
Number of creatinine, AST/ALT | 4 weeks
  Creatinine in mg/dl, AST/ALT in UL

CONTACTS AND LOCATIONS:
Overall Officials: Youngmin Ye, Dr, Study Director — Ajou University
Locations (1):
- Ajou University Medical Hospital, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No